CLINICAL TRIAL: NCT03226808
Title: Post Market Clinical Follow-up Study of the Zimmer Vivacit-E Highly Crosslinked Polyethylene Liner Used With the Continuum Acetabular Shell
Brief Title: Vivacit-E Post-market Follow-up Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMU2011-09H
Record Dates: First submitted 2016-08-11; First posted 2017-07-24 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis; Avascular Necrosis of Bone of Hip; Post-traumatic; Arthrosis; Congenital Hip Dysplasia
MeSH Terms: conditions — Osteoarthritis; Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vivacit-E Liner (Other): All subjects enrolled receive the study implant.
  Interventions: Device: Vivacit-E Liner

INTERVENTIONS:
Device: Vivacit-E Liner — All subjects enrolled will receive the Vivacit-E liner.

SUMMARY:
The objectives of this study are to obtain clinical performance (outcomes) data and survivorship for commercially available Vivacit-E (HXPE) liners. This will be done by analysis of polyethylene wear, validated outcome measurement tools, radiographs, and reported adverse events data.

DETAILED DESCRIPTION:
Safety will be evaluated by monitoring the frequency and incidence of adverse events.

Performance will be determined by assessment of the overall pain and functional performances, survivorship, health status and radiographic parameters of all enrolled study subjects who receive the Vivacit-E HXPE Liner with the Continuum acetabular shell.

In addition, the implanted Vivacit-E HXPE Liners will be evaluated for bedding in, and linear and volumetric wear by the Martell 2-D method at 6 weeks and 1, 2, 4, & 5 years postoperatively.

Pain and functional performance will be measured using the Harris Hip and High Activity Arthroplasty Scores. Survivorship will be based on removal or intended removal of the device and through analysis of radiographs, and health status will be determined by evaluation of the EQ-5D.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 60 years of age, inclusive.
* Patient is skeletally mature.
* Patient qualifies for primary unilateral or bilateral total hip arthroplasty (THA) based on physical exam and medical history including at least one of the following:
* Osteoarthritis
* Avascular necrosis (AVN)
* Post-traumatic arthritis
* Congenital hip dysplasia
* Patient has no history of previous total hip replacement or arthrodesis of the affected hip joint(s).
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the IRB/EC approved informed consent.

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient has a total prosthetic hip replacement device (including surface replacement arthroplasty, endoprosthesis, etc. in the affected hip joint(s).
* Inflammatory Arthritis
* Rheumatoid Arthritis
* The patient is:

  * a prisoner mentally incompetent or unable to understand what participation in the study entails a known alcohol or drug abuser
  * anticipated to be non-compliant
  * The patient has an acute, chronic, or systemic infection(s).
  * The patient has total or partial absence of the muscular or ligamentous apparatus.
  * The patient has neuromuscular compromise, vascular deficiency or other conditions in the affected limb that may lead to inadequate skeletal fixation.
  * The patient has osteoradionecrosis.
  * The patient has lack of bony structures proximal or distal to the operative joint, so that good implant fixation is unlikely or impossible.
  * The patient has local bone tumors/cysts in the bone to be retained that the implanting surgeon determines could inhibit implant fixation.
  * The patient is skeletally immature.
  * The patient has any concomitant disease that can jeopardize the functioning and the success of the implant.
  * The patient is known to be pregnant.
  * The patient has a known sensitivity or allergic reaction to one or more of the implanted materials which include metal (titanium, tivanium, tantalum, cobalt, chromium, nickel) and ceramic.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival of the study device; whether or not it is still implanted in the subject | 10 years
  Survival is classified as removal of the study device for any reason

SECONDARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (safety) | 10 years
  Safety is assessed by monitoring the frequency and incidence of all adverse events, with particular focus on those that may be related to the study device.
Harris Hip Score | 10 years
  Functional outcomes are measured with the Harris Hip Score, including range of motion, pain level, activity levels and patient satisfaction.
Patient activity level | 10 years
  Patient activity level is assessed with the High Activity Arthroplasty score, filled out by the patient.
Patient Quality of Life | 10 years
  This is another self-assessment by means of the EQ-5D score, which measures the patient's perceived quality of life.
Radiographic analysis | 2 years
  Patient x-rays will undergo a Martell analysis by Dr. John Martell to evaluate radiolucencies, osteolysis, sbusidence, cup migration and polyethylene wear.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Boylan, MBA, Study Director — Zimmer Biomet
Locations (5):
- United States (5):
  - Denver Hip and Knee, Inc., Parker, Colorado
  - Department of Orthopaedics University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Rothman Institute, Philadelphia, Pennsylvania
  - Texas Institute for Hip and Knee Surgery, Austin, Texas

IPD SHARING:
Plan to Share IPD: No